CLINICAL TRIAL: NCT02669927
Title: Frailty and Postoperative Shock
Status: Completed | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Forget Patrice, PI, Université Catholique de Louvain
Other Study IDs: 2012/17DEC/539
Record Dates: First submitted 2016-01-27; First posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Frailty; Elderly
Keywords: hip surgery; frail older people
MeSH Terms: conditions — Frailty | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Observational

SUMMARY:
To find an objective, affordable and manageable way to measure frailty in elderly patients and to examine relationship between peri-operative metabolism of frail older people and outcome after hip surgery.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized in St-Luc Hospital (Belgium) for hip surgery between 2013 and 2015

Exclusion Criteria:

* non-traumatic hip fracture
* refusal

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 53 patients (age = 82 ans [56-98]) hospitalized in St-Luc Hospital (Belgium) for hip surgery between 2013 and 2015
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Mortality | up to one year